CLINICAL TRIAL: NCT05431452
Title: Evaluation of the Effect of Fetal Position, Kangaroo Care, Breast Milk and Combined Fetal Position and Kangaroo Care in Reducing Pain During Heel Blood Collection in Preterm Newborns.
Brief Title: Reducing Pain During Heel Blood Collection in Preterm Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Serife Tutar, Assistant professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 206337
Record Dates: First submitted 2022-04-21; First posted 2022-06-24 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Preterm Birth; Pain, Acute
Keywords: preterm birth; pain; nursing care
MeSH Terms: conditions — Premature Birth; Acute Pain; Pain | interventions — Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Control Group) (No Intervention): There is no non-pharmacological method applied during routine heel blood collection in the clinic where the research will be conducted. No intervention will be applied to this group within the scope of the research. In order to minimize the risk of aspiration during the procedure, the head of the bed in the incubator will be elevated at a 45-degree angle. The 1st minute before the procedure, the 1st minute and the 2nd minute during and after the procedure will be recorded with a video camera and the data on the monitor will be recorded in the "Physiological Parameters Measurement Form".
- Group 2 (Breast milk) (Experimental): 2 minutes before the procedure, the bedside of the baby will be raised at an angle of 45 degrees and 2 ml of breast milk will be given by the research clinic nurse with the help of a sterile injector, provided that each baby will be their own breast milk. Heel blood collection will be performed 2 minutes after breast milk is given. The 1st minute before the procedure, the 1st and 2nd minutes during and after the procedure will be recorded with a video camera and the data on the monitor will be recorded in the "Physiological Parameters Measurement Form".
  Interventions: Other: Pain management
- Group 3 (Supine Fetal Position) (Experimental): This method is a lower form of the method of taking the baby into the nest and is defined as the process of keeping the baby's upper and lower extremities flexed by hand, and taking the body into a closed position close to the midline. While applying this method, the baby can be placed in a lateral, supine or prone position (Neto et al., 2020).
  In our research, according to the literature, the baby will be placed in the fetal position 3 minutes before the procedure, and the baby will be kept in the fetal position for 3 minutes after the procedure. The 1st minute before the procedure, the 1st and 2nd minutes during and after the procedure will be recorded with a video camera and the data on the monitor will be recorded in the "Physiological Parameters Measurement Form".
  Interventions: Other: Pain management
- Group 4 (Kangaroo maternal care) (Experimental): 10 minutes before the procedure, the mother will be placed on the mother's chest at an angle of 60 degrees, with only the diaper left under the baby in the baby adjustment room, in a way that it will contact the mother's chest directly from skin to skin. In order not to lower the newborn's body temperature, a thin blanket will be covered on his back and the mother will be asked to gently soothe the baby's movements by wrapping her hands around the newborn's back. The mother will be instructed not to make additional movements such as stroking, talking, feeding and shaking her baby. After 10 minutes of kangaroo mother care, heel blood collection will be performed and after the procedure, kangaroo mother care will continue for 2 more minutes. The 1st minute before the procedure, the 1st and 2nd minutes during and after the procedure will be recorded with a video camera and the data on the monitor will be recorded in the "Physiological Parameters Measurement Form".
  Interventions: Other: Pain management
- Group 5 (Supine Fetal position + Breast milk) (Experimental): The head of the baby's bed is elevated to a 45-degree angle and before the procedure, 2 ml of breast milk will be given with the help of a sterile injector by the research clinical nurse, on the condition that each baby has its own breast milk, and then the baby will be placed in the fetal position (Shah et al., 2012; Shukla et al. , 2018). After the baby is held in the fetal position for 3 minutes, heel blood sampling will be performed. The 1st minute before the procedure, the 1st and 2nd minutes during and after the procedure will be recorded with a video camera and the data on the monitor will be recorded in the "Physiological Parameters Measurement Form". In line with the literature recommendations, the baby will be supported in the fetal position for 3 minutes after the procedure (Axelin et al. 2006; Cignacco et al. 2010; Obeidat et al. 2009; Çağlayan and Balci, 2014).
  Interventions: Other: Pain management
- Group 6 (Kangaroo care + Breast milk) (Experimental): The head of the baby's bed will be raised at an angle of 45 degrees and before the procedure, 2 ml of breast milk will be given by the research clinical nurse with the help of a sterile injector, provided that each baby is breast milk, and then the mother will be in direct skin-to-skin contact with the mother's breast, with only the diaper under the baby in the baby adaptation room. It will be placed on the mother's chest at an angle of 60 degrees. The mother will be instructed not to make additional movements such as stroking, talking, feeding and shaking her baby. After 10 minutes of kangaroo mother care, heel blood collection will be performed and after the procedure, kangaroo mother care will continue for 2 more minutes. The 1st minute before the procedure, the 1st and 2nd minutes during and after the procedure will be recorded with a video camera and the data on the monitor will be recorded in the "Physiological Parameters Measurement Form".
  Interventions: Other: Pain management

INTERVENTIONS:
Other: Pain management — Nonpharmacological pain management during blood collection in preterm infants
  Arms: Group 2 (Breast milk); Group 3 (Supine Fetal Position); Group 4 (Kangaroo maternal care); Group 5 (Supine Fetal position + Breast milk); Group 6 (Kangaroo care + Breast milk)

SUMMARY:
Pharmacological and non-pharmacological methods are used to control interventional pain in preterm newborns. Non-pharmacological methods should be preferred in the management of pain, especially during painful minor invasive procedures (blood collection, orogastric tube insertion, aspiration, etc.) applied during the day. Some of these methods are; kangaroo care, breast milk, fetal positioning, breastfeeding, listening to music and massage.

Taking heel blood from babies who are being treated in the neonatal intensive care unit is among the duties, authorities and responsibilities of neonatal intensive care nurses. In addition, the effective management of pain by using non-pharmacological methods is among the professional ethical responsibilities of nurses working in neonatal intensive care units. While fulfilling these responsibilities, nurses should conduct researches with high levels of evidence and benefit from the researches effectively. In this context, determining the most effective non-pharmacological method and activating it in a clinical setting form the basis of nursing practices. In this context, the aim of our research is; The aim of this study is to evaluate the effects of fetal position, kangaroo care, combined fetal position with breast milk and breast milk, and kangaroo care in reducing pain during heel blood collection in preterm newborns.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of fetal position, kangaroo care, combined fetal position with breast milk and breast milk, and kangaroo care in reducing pain during heel blood collection in preterm newborns. The sample of the study will consist of late preterm newborns who meet the inclusion criteria of the study. It is envisaged that 40 babies will be included in the sample for each group. Randomization will be done in order to provide an equal number of samples for the intervention and control groups in the study. In the randomization to be made, the "simple randomization method" will be used in order to provide equal samples for all three groups. The data of the study will be collected by the clinical nurse working as a nurse in the clinic where the research is conducted, in accordance with the randomization scheme. Physiological parameters of all babies will be monitored on the monitor during the interventions. During the research, all groups will be video-recorded for 10 minutes before the procedure, during the procedure and for 5 minutes after the procedure. After the data of the study are collected, all video recordings will be examined by two researchers (a neonatal intensive care nurse and a neonatal intensive care specialist) and PIPP-R The scale will be filled in by these two independent observers. Descriptive statistics (mean, standard deviation) will be used for the quantitative variables of the research determined by measurement, and descriptive statistics (number, percentage) will be used for the qualitative variables determined by counting. The conformity of the data to be used with the normal distribution will be determined by the Shapiro-Wilk test. In paired comparisons between variables with two categories such as gender, t-test, Analysis of Variance will be applied to find the differences between variables with three or more categories such as group. Paired-sample t-test will be applied between dependent groups for the features that are significant as a result of the analysis of variance. Mann Whitney U test, Wilcoxon test and correlation analyzes will be used to evaluate the relationships between dependent and independent variables. Results will be evaluated at 95% confidence interval and p<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Gestation week between 34(0)/7 - 36(6)/7 weeks
* Stable physiological condition
* Able to maintain spontaneous breathing
* Able to take breast milk
* Not exposed to a painful procedure at least half an hour before the intervention.
* Late preterm newborns not taking opioid or non-opioid analgesics will be included in the -study.

Exclusion Criteria:

* Receiving mechanical ventilator support
* Congenital anomaly
* Using analgesic/narcotic analgesic drugs
* Babies who receive treatment with continuous sedation will not be included in the study.

Ages: 3 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain management | 10 month
  Management of pain heel puncture in premature newborn. The parameter for pain management will be determined by the Premature Infant Pain Profile (PIPP)

CONTACTS AND LOCATIONS:
Overall Officials: Şerife Tutar, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to publish the research data in the form of an article.